CLINICAL TRIAL: NCT05581524
Title: V.A.S.C. (Vacuum Assisted Sclerotherapy Performed by Catheter)
Brief Title: Vacuum Assisted Sclerotherapy Performed by Catheter
Acronym: VASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I-VASC S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPS01
Record Dates: First submitted 2022-10-05; First posted 2022-10-14 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-03

CONDITIONS: Varicose Veins of Lower Limb
Keywords: varicose veins; empty-vein sclerotherapy; chemical ablation; venous catheter
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Intervention Model Description: V.A.S.C. is a multicentric, prospective, open label, non-randomized PMCF study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VELEX (Experimental): Treatment of varicose veins of lower limbs by means of chemical ablation or empty-vein sclerotherapy
  Interventions: Device: VASC

INTERVENTIONS:
Device: VASC — At day 0 the patient will undergo the VASC treatment procedure with VelexTM device. VelexTM venous catheter is inserted in the introducer and pushed in the desired position under echo guidance. At 7 days, 1, 3 and 6 months after the procedure, the patients will undergo a clinical examination and an echo-color doppler assessment.
  Other Names: Velex

SUMMARY:
VelexTM Venous Catheter is a venous catheter for temporary use to treat a vein isolated segment, designed for the treatment of varicose veins of lower limbs by means of chemical ablation or empty-vein sclerotherapy.

V.A.S.C. is a multicentric, prospective, open label, non-randomized PMCF study of VelexTM venous catheter used according to the indication of use within the scope of the CE mark.

VelexTM venous catheter is intended for patients with varicose veins of lower limbs. The total minimum number of patients is 24 and the maximum 36 for the two centers participating. Each center shall enroll at least 8 patients andno more than 28.

DETAILED DESCRIPTION:
V.A.S.C. is a multicentric prospective, open label, non-randomized PMCF study of VelexTM venous catheter for patients with varicose veins of lower limb.

The study is designed as a post-market clinical follow-up, aimed at collecting clinical data of VelexTM venous catheter used according to the indication of use within the scope of the CE mark.

The study will enrol a maximum number of 36 patients at the participating sites. All the subjects will be evaluated at immediate post-procedure, 7 days, 1, 3 and 6 months after the procedure.

The eligibility criteria are compliant with the indication of use within the scope of the CE mark.

Several preclinical tests were carried out for assessing the safety of VelexTM venous catheter: in vitro tests, biocompatibility and preclinical-vivo test.

In-vitro test All the in-vitro tests were performed on samples at time zero and after aging, in order to simulate conditions of transport and storage of the device Biocompatibility The biocompatibility assessment included the overall evaluation of the device, including the manufacturing materials of the various components, the manufacturing processes, the clinical use of the device, including the expected anatomical location, and the frequency and duration of exposure.

According to ISO 10993-1, VelexTM venous catheter is classified as an external communication device with limited contact duration (≤24 hours), with contact with circulating blood. According to this category, dedicated tests were performed to provide data regarding specific biological effects:

* Cytotoxicity
* Sensitization
* Irritation or intracutaneous reactivity
* Pyrogenicity
* Acute systemic toxicity
* Hemocompatibility In all the biocompatibility test, the samples met the acceptance criteria. On the basis of biocompatibility tests carried out, VelexTM venous catheter device complies with the biocompatibility requirements according to ISO 10993-1: 2018.

Preclinical in-vivo test A preclinical in-vivo test was performed on ovine animal model in order to evaluate the safety of the device in conditions consistent with the clinical use and to verify the echogenicity of the device under ultrasound. Sclerotherapy procedure was simulated in jugular vein of adult sheep.

Most of the procedures (9/15) were successfully completed. Among the remaining 6 cases, 4 cases resulted in an incomplete procedure due to out of procedure (not conform to the IFU); in 2 procedures with the same catheter the user encountered resistance to catheter movement, therefore the catheter was retrieved but no damage to the device or to the vein was detected.

In order to simulate the dynamic method, the catheter with inflated balloons was repeatedly moved along the vessel without any issue.

By means of diagnostic imaging, the position of the catheter was checked, as well as balloons inflation and deflation, confirming the safety of the mechanism of action of the device. Hereafter, the device features positively assessed by these tests are listed:

* Safe compatibility with Seldinger technique;
* Good pushability/trackability;
* Excellent echogenicity;
* Safe inflation/deflation of balloons;
* Safe isolation of vein segment;
* Safe fluid injection;
* Safe displacement of the catheter;
* Safe fluid aspiration;
* Safe retrieval of the catheter;
* Safe synchronism mechanism (handle). In addition, it is remarkable that no damages to the vein nor to catheter were observed. Damages to catheter were observed only when out of procedures occurred.

The in-vivo test confirmed the results of the in-vitro test in term of safety and ease of use of VelexTM venous catheter.

Evaluation of clinical data that are relevant to the proposed clinical investigation At the moment, the clinical evaluation of VelexTM catheter is based on literature data regarding the use of catheters for sclerotherapy.

Sclerotherapy is a well established treatment for small varicose vein but there are some limitations due to lack of standardization of the technique and the anatomical recurrence rate remains higher than the other endovenous options. The use of long catheters for sclerotherapy has been described since 1997. Through the use of catheters with occlusion balloons, the sclerosing agent can be maintained in contact with the venous inner wall for the period necessary to stimulate an endothelial response; furthermore, the occlusion balloon decreases the probability of damage to the structures of the deep venous system due to the migration of the sclerosant.

The major challenge that remains with any type of catheter is how to standardize the dose of therapeutic agent to be used during the procedure and to be able to distribute it evenly along the vascular wall.

Clinical data from scientific literature show that sclerotherapy with a catheter under echo guidance is safe and leads to clinical benefit for patients. The use of VelexTM is consistent with the current medical knowledge in the treatment of varicose veins. Indeed, VelexTM is a catheter with features that allow to control the concentration of sclerosant agent in an isolated venous segment emptied from blood and to keep it in place for the time deemed necessary.

VelexTM Venous Catheter is a venous catheter for temporary use to treat a vein isolated segment, designed for the treatment of varicose veins of lower limbs by means of chemical ablation or empty-vein sclerotherapy.

The device allows to isolate the vein section to be treated, to release the sclerosant agent in the lesion to be treated through the medication administration holes and to recapture the injected liquid, preventing undesired side effects.

It is composed by the following parts:

* Three-balloon catheter: main body and invasive part of the device;
* Handle: it manages the balloon and the medication infusion;
* Syringe preparation lines: silicone tubes to be connected to the handle in order to fill the syringes;
* Depth marker: sliders (C-shape rings) connected by a spacer. VelexTM venous catheter is intended to temporary inhibit blood flow in isolated sections of the peripheral veins of the lower limbs to infuse therapeutic agents (foam excluded) prescribed by physician for sclerotherapy.

The intended purpose of VelexTM venous catheter in the PMCF study coincides with the indication of use within the scope of the CE mark.

VelexTM venous catheter is intended for patients affected by lower limb CVD. The suitability of the patient is to be verified case by case by the specialized physician, by means of proper physical examination and evaluation of superficial and deep venous system by means of color Doppler echocardiography.

VelexTM venous catheter should be used by physicians having a deep knowledge of:

* vascular anatomy
* venous system pathology
* endovascular peripheral procedures and endovascular methods
* Seldinger technique or techniques for surgical isolation of a superficial vein
* diagnostic methods, especially peripheral echo color Doppler echocardiography of deep and superficial venous system and angiography.

VelexTM venous catheter shall be inserted in a vein of the lower limb by means of direct phlebotomy or Seldinger technique with 7 Fr introducer, and placed in the desired position under echo guidance.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old
* Weight >45 kg
* Asymptomatic or presence of at least one of the following symptoms: pain, heaviness, tiredness, itching, night cramps, restlessness, general discomfort, swelling.
* GSV standing diameter between 4 and 12 mm along the whole veins (measured by Duplex ultrasound)
* Willingness to undergo follow-up visits
* Ability to understand scope, content and risks of the study, and provide informed consent to participation

Exclusion Criteria:

* Contraindications for endovascular procedures (fever, infectious processes, tumor diseases, hemorragic diathesis)
* Any disease or condition contraindicating sclerotherapy treatment
* Peripheral symptomatic arterial pathology (ankle brachial index ABI <0.80)
* History or suspect of Deep Venous Thrombosis (DVT) or Superficial Venous Thrombosis of Great Saphenous Vein (SVT of GSV)
* GSV standing diameter > 12 mm for vein segments longer than 3 cm or diameter < 4 mm for segments longer than 5 cm
* Caprini score >10
* Pregnancy and breastfeeding
* Previous treatments of venous pathologies in the leg (excluding telangiectasis and reticular venulas)
* Allergy to sclerosant agent
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Confirm the safety and performances of VelexTM device when used in accordance with the Instructions for Use | 3 months
  After 3 months, patients will be asked to fill a questionnaire of quality of life.
Pain level | At day 0 (day of procedure)
  Evaluated and recorded the pain during the procedure with the pain score scale:
  Visual analogue scale (VAS) 0= NO PAIN 1-3=MILD PAIN 4-6= MODERATE/SEVERE PAIN 7-9= VERY SEVERE PAIN 10=WORST PAIN POSSIBLE
Pain level | 7 days from the procedure
  Evaluated and recorded the pain post the procedure with the pain score scale:
  Visual analogue scale (VAS) 0= NO PAIN 1-3=MILD PAIN 4-6= MODERATE/SEVERE PAIN 7-9= VERY SEVERE PAIN 10=WORST PAIN POSSIBLE

CONTACTS AND LOCATIONS:
Overall Officials: Mario MS Salerno, Study Chair — I-VASC S.r.l
Locations (2):
- Italy (2):
  - IRCCS Policlinico San Donato, Milan, Milan
  - IRCCS San Raffaele, Milan, Milan